CLINICAL TRIAL: NCT02774343
Title: PPARγ Agonist Treatment for Cocaine Dependence
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Joy Schmitz, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-12-0421; P50DA009262 (NIH)
Record Dates: First submitted 2016-05-06; First posted 2016-05-17 (Estimated); Results first posted 2018-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-03

CONDITIONS: Cocaine Use Disorder; Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Pioglitazone; Starch; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone + Therapy + Contingency Management (Experimental): Subjects randomized to pioglitazone begin with a starting dose of 15 mg daily administered. The dose will be titrated up to 30mg on the second week and 45 mg on the third week of the study. Subjects will remain on 45 mg of pioglitazone until the end of week 12. At the end of week 12 the study medication will be discontinued.
  Interventions: Drug: Pioglitazone; Behavioral: Therapy; Behavioral: Contingency Management
- Placebo + Therapy + Contingency Management (Placebo Comparator): Subjects randomized to placebo receive placebo capsules once daily across all twelve weeks of the study.
  Interventions: Drug: Placebo; Behavioral: Therapy; Behavioral: Contingency Management

INTERVENTIONS:
Drug: Pioglitazone — Subjects randomized to pioglitazone begin with a starting dose of 15 mg daily administered. The dose will be titrated up to 30mg on the second week and 45 mg on the third week of the study. Subjects will remain on 45 mg of pioglitazone until the end of week 12. At the end of week 12 the study medication will be discontinued.
  Other Names: Actos
  Arms: Pioglitazone + Therapy + Contingency Management
Drug: Placebo — Subjects randomized to placebo receive placebo capsules once daily across all twelve weeks of the study.
  Other Names: corn starch
  Arms: Placebo + Therapy + Contingency Management
Behavioral: Therapy — Cognitive-behavioral therapy 1 hour per week
Behavioral: Contingency Management — Prize-based contingency management for attendance

SUMMARY:
The purpose of this research study is to determine whether a medication called pioglitazone (trade name Actos) can reduce behavioral problems associated with cocaine use, improve brain structural changes associated with cocaine use and reduce cocaine craving and drug use in cocaine dependent patients.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for cocaine dependence
* At least one cocaine positive urine during screening
* Female subjects: a negative pregnancy test
* Be in acceptable health on the basis of interview, medical history and physical exam
* Be able to understand the consent form and provide written informed consent
* Be able to provide the names of at least 2 persons who can generally locate their whereabouts.

Exclusion Criteria:

* Current Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV diagnosis of any psychoactive substance dependence other than cocaine marijuana, alcohol, or nicotine
* Any serious medical or psychiatric illness and/or clinically significant abnormal laboratory value, which in the judgment of the Principal Investigator or his/her designee would make study participation unsafe, or would make treatment compliance difficult or put the study staff at undue risk
* Significant current suicidal or homicidal ideation
* Medical conditions contraindicating pioglitazone pharmacotherapy (e.g., congestive heart failure as determined by Framingham criteria, clinically significant edema, clinically significant liver disease, hypoglycemia, diabetes, history of bladder cancer)
* Taking medications known to have significant drug interactions with the study medication (CYP2C8 inhibitors or inducers, antihyperglycemic medications)
* Currently being treated for substance misuse with medication
* Conditions of probation or parole requiring reports of drug use to officers of the court
* Impending incarceration
* Pregnant or planning to become pregnant during the course of the trial or nursing for female patients
* Inability to read, write, or speak English (many of the research instruments in this study only exist in English)
* Having plans to leave the immediate geographical area within 3 months
* Unwillingness to sign a written informed consent form
* Unwillingness to use a barrier method of birth control during the study for female patients
* History of pacemaker or metal implants or welding or metal work without protective eyewear (for risk of MRI scans).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joy M Schmitz, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pioglitazone + Therapy + Contingency Management | Placebo + Therapy + Contingency Management
Started | 15 | 15
Received at Least One Capsule | 12 | 14
Completed | 9 | 12
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone + Therapy + Contingency Management | Placebo + Therapy + Contingency Management | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (7.1) | 47.4 (7.8) | 47.8 (7.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 11 | 11 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Craving as Assessed by the Brief Substance Craving Scale (BSCS)
Description: The brief substance craving scale (BSCS) is a 16-item, self-report instrument assesses craving for cocaine and other substances of abuse over a 24 hour period. The domains of intensity, frequency, and duration are recorded on a five-point Likert scale. The range of scores for each domain is 0 to 4, and the total score is the sum of all three domains. The total score range is 0 to 12, and higher scores indicate higher craving (worse outcome.)
Time Frame: Baseline, week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11, week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pioglitazone + Therapy + Contingency Management | Placebo + Therapy + Contingency Management
Number analyzed (Participants) | 12 | 14
units on a scale
  baseline | 5.57 (2.47) | 6.23 (3.30)
  week 1 | 5.00 (3.36) | 5.08 (3.06)
  week 2 | 4.42 (2.11) | 2.91 (2.55)
  week 3 | 4.00 (3.33) | 3.82 (3.89)
  week 4 | 4.00 (3.16) | 3.18 (2.75)
  week 5 | 2.60 (2.55) | 3.82 (2.79)
  week 6 | 3.22 (2.78) | 3.45 (3.39)
  week 7 | 2.12 (1.64) | 4.36 (3.14)
  week 8 | 3.25 (2.12) | 3.55 (2.38)
  week 9 | 2.88 (2.53) | 3.82 (3.25)
  week 10 | 2.56 (2.55) | 3.36 (2.98)
  week 11 | 2.89 (2.62) | 3.82 (2.56)
  week 12 | 2.00 (2.39) | 3.55 (2.88)

2. Primary Outcome: Craving as Assessed by the Obsessive Compulsive Drug Use Scale (OCDUS)
Description: The obsessive compulsive drug use scale (OCDUS) measures the level of craving for cocaine during the past week. The mean score over all time points is reported in this outcome measure (i.e., a summary score is reported). The scale was administered once weekly. It consists of 12 items. The score range is 0 to 60, and higher scores indicates greater craving.
Time Frame: Weeks 1-12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pioglitazone + Therapy + Contingency Management | Placebo + Therapy + Contingency Management
Number analyzed (Participants) | 12 | 14
units on a scale | 19.1 (3.5) | 21.36 (8.7)

3. Primary Outcome: Cue Reactivity as Assessed by a Visual Analogue Scale (VAS) of Cocaine Craving
Description: Every two weeks, visual analog scale ratings of craving (VAS craving) consisting of 100 mm line, anchored by 0 "not at all" and 100 "extremely," were used to assess cocaine craving right now, craving on average in the past week, and the worst craving in the past week. Data were analyzed as a total score, which is the sum of the scores for the three questions.
Time Frame: Baseline, week 2, week 4, week 6, week 8, week 10, week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pioglitazone + Therapy + Contingency Management | Placebo + Therapy + Contingency Management
Number analyzed (Participants) | 12 | 14
units on a scale
  baseline | 57.50 (22.83) | 52.29 (29.49)
  week 2 | 53.76 (23.10) | 40.31 (29.38)
  week 4 | 37.93 (22.30) | 35.58 (29.00)
  week 6 | 21.75 (22.97) | 29.86 (31.27)
  week 8 | 25.70 (23.34) | 35.88 (34.20)
  week 10 | 18.33 (24.38) | 31.42 (35.61)
  week 12 | 15.38 (28.91) | 27.86 (30.20)

4. Primary Outcome: Brain White Matter (WM) Integrity as Assessed by Diffusion Tensor Imaging (DTI) Fractional Anisotropy (FA) Value (Region - Posterior Thalamic Radiation)
Description: DTI scans were acquired on a Philips Integra 3T magnet. Fractional anisotropy (FA) is a summary measure of the integrity of white matter neurons that provides a dimensionless index of the expected movement of water molecules inside and across the neuron. Higher values of FA indicate better neuronal integrity (that is, less movement of water across the neuron). There is no range of values, as this is a dimensionless index.
Time Frame: Baseline and Week 12
Population: Although 21 completed the study, only 18 were analyzed for this measure. This is because DTI FA data was collected for only 18 subjects. Reasons for not completing DTI: 1 subject had a brain abnormality; 1 subject refused to do the scan; and 1 scan was not completed due to scanner shutdown for maintenance.
Measure: Mean (Standard Deviation); unit: DTI Fractional Anisotropy (FA) value
Arm/Group | Pioglitazone + Therapy + Contingency Management | Placebo + Therapy + Contingency Management
Number analyzed (Participants) | 8 | 10
DTI Fractional Anisotropy (FA) value
  baseline | 542.27 (24.60) | 546.26 (27.02)
  week 12 | 546.84 (32.79) | 535.14 (27.61)

5. Primary Outcome: Brain White Matter (WM) Integrity as Assessed by Diffusion Tensor Imaging (DTI) Fractional Anisotropy (FA) Value (Region - Anterior Thalamic Radiation)
Description: as for outcome 4
Time Frame: Baseline and Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: DTI Fractional Anisotropy (FA) value
Arm/Group | Pioglitazone + Therapy + Contingency Management | Placebo + Therapy + Contingency Management
Number analyzed (Participants) | 8 | 10
DTI Fractional Anisotropy (FA) value
  baseline | 518.20 (24.42) | 530.31 (26.28)
  week 12 | 522.40 (30.85) | 523.00 (36.46)

6. Primary Outcome: Brain White Matter (WM) Integrity as Assessed by Diffusion Tensor Imaging (DTI) Fractional Anisotropy (FA) Value (Region - Splenium of Corpus Callosum)
Description: as for outcome 4
Time Frame: Baseline and Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: DTI Fractional Anisotropy (FA) value
Arm/Group | Pioglitazone + Therapy + Contingency Management | Placebo + Therapy + Contingency Management
Number analyzed (Participants) | 8 | 10
DTI Fractional Anisotropy (FA) value
  baseline | 645.49 (48.82) | 635.81 (26.26)
  week 12 | 655.41 (26.73) | 620.98 (35.51)

7. Primary Outcome: Brain White Matter (WM) Integrity as Assessed by Diffusion Tensor Imaging (DTI) Fractional Anisotropy (FA) Value (Region - Genu of Corpus Callosum)
Description: as for outcome 4
Time Frame: Baseline and Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: DTI Fractional Anisotropy (FA) value
Arm/Group | Pioglitazone + Therapy + Contingency Management | Placebo + Therapy + Contingency Management
Number analyzed (Participants) | 8 | 10
DTI Fractional Anisotropy (FA) value
  baseline | 566.66 (44.18) | 562.52 (29.34)
  week 12 | 575.06 (30.78) | 547.15 (37.45)

8. Primary Outcome: Brain White Matter (WM) Integrity as Assessed by Diffusion Tensor Imaging (DTI) Fractional Anisotropy (FA) Value (Region - External Capsule)
Description: as for outcome 4
Time Frame: Baseline and Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: DTI Fractional Anisotropy (FA) value
Arm/Group | Pioglitazone + Therapy + Contingency Management | Placebo + Therapy + Contingency Management
Number analyzed (Participants) | 8 | 10
DTI Fractional Anisotropy (FA) value
  baseline | 420.68 (22.35) | 418.71 (15.92)
  week 12 | 423.91 (17.23) | 418.25 (16.98)

9. Primary Outcome: Brain White Matter (WM) Integrity as Assessed by Diffusion Tensor Imaging (DTI) Fractional Anisotropy (FA) Value (Region - Cingulum)
Description: as for outcome 4
Time Frame: Baseline and Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: DTI Fractional Anisotropy (FA) value
Arm/Group | Pioglitazone + Therapy + Contingency Management | Placebo + Therapy + Contingency Management
Number analyzed (Participants) | 8 | 10
DTI Fractional Anisotropy (FA) value
  baseline | 465.06 (22.35) | 463.91 (15.92)
  week 12 | 471.40 (17.23) | 465.75 (16.98)

10. Secondary Outcome: Feasibility - Subject Retention as Assessed by Number of Participants Who Completed All 12 Weeks of the Study
Time Frame: week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Pioglitazone + Therapy + Contingency Management | Placebo + Therapy + Contingency Management
Number analyzed (Participants) | 15 | 15
Participants | 12 | 11

11. Secondary Outcome: Feasibility - Medication Compliance as Assessed by Percentage of Urine Samples That Were Riboflavin-Positive
Description: Riboflavin was added to pill capsules as a marker of medication compliance. The percentage over all time points is reported in this outcome measure. Urine samples were collected once weekly.
Time Frame: weeks 1 - 12
Measure: Mean (Standard Error); unit: percentage of urine samples
Arm/Group | Pioglitazone + Therapy + Contingency Management | Placebo + Therapy + Contingency Management
Number analyzed (Participants) | 12 | 14
percentage of urine samples | 96.2 (0.055194) | 95.4 (0.055987)

12. Secondary Outcome: Feasibility - Medication Compliance as Assessed by Percentage of Self-reports That Indicate Capsules Were Taken
Description: A modified Timeline Followback (TLFB) procedure was used for self-reports. The percentage over all time points is reported in this outcome measure. Self-reports were collected once weekly.
Time Frame: weeks 1 - 12
Measure: Mean (Standard Error); unit: percentage of self-reports
Arm/Group | Pioglitazone + Therapy + Contingency Management | Placebo + Therapy + Contingency Management
Number analyzed (Participants) | 12 | 14
percentage of self-reports | 84.1 (0.105562) | 86.9 (0.090174)

13. Secondary Outcome: Feasibility - Tolerability as Assessed by Number of Participants Reporting Side Effects
Time Frame: week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Pioglitazone + Therapy + Contingency Management | Placebo + Therapy + Contingency Management
Number analyzed (Participants) | 12 | 14
Participants
  drowsiness | 0 | 1
  not sleeping well | 2 | 1
  headache | 0 | 1
  nervousness | 0 | 2
  blurry vision | 0 | 2
  dizziness | 0 | 1
  nausea | 0 | 1
  vomiting | 1 | 1
  diarrhea | 2 | 1
  stomach pain | 3 | 2
  muscle aches | 0 | 1
  shortness of breath | 0 | 1
  cough | 4 | 1
  increased urination | 4 | 1
  change in sexual function | 1 | 1
  weakness | 0 | 1
  fatigue | 1 | 0
  difficulty walking | 1 | 0
  fever or chills | 0 | 2
  loss of appetite | 0 | 1
  confusion | 0 | 1
  cloudiness | 0 | 1
  memory loss | 1 | 0

14. Secondary Outcome: Feasibility - Tolerability as Assessed by Number of Participants With Serious Adverse Events
Time Frame: week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Pioglitazone + Therapy + Contingency Management | Placebo + Therapy + Contingency Management
Number analyzed (Participants) | 12 | 14
Participants | 0 | 0

15. Secondary Outcome: Cocaine Use as Assessed by Percentage of Urine Samples That Were Cocaine-positive
Description: The mean percentage over all time points is reported in this outcome measure. Urine samples were collected once weekly.
Time Frame: Weeks 1-12
Measure: Mean (Standard Deviation); unit: percentage of urine samples
Arm/Group | Pioglitazone + Therapy + Contingency Management | Placebo + Therapy + Contingency Management
Number analyzed (Participants) | 12 | 14
percentage of urine samples | 44 (0.34) | 50 (0.4)

16. Secondary Outcome: Cocaine Use as Assessed by Percentage of Self-reports That Indicate Cocaine Use
Description: A modified Timeline Followback (TLFB) procedure was used to assess cocaine use. The mean percentage over all time points is reported in this outcome measure. Self-reports were collected once weekly.
Time Frame: Weeks 1-12
Measure: Mean (Standard Deviation); unit: percentage of self-reports
Arm/Group | Pioglitazone + Therapy + Contingency Management | Placebo + Therapy + Contingency Management
Number analyzed (Participants) | 12 | 14
percentage of self-reports | 35 (0.3) | 29 (0.28)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Side effects are listed in Outcome Measure 13 are side effects; however, side effects were not considered to be adverse events.
Arm/Group | Pioglitazone + Therapy + Contingency Management | Placebo + Therapy + Contingency Management
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 0/12 | 0/14

LIMITATIONS AND CAVEATS:
Small sample size; restricted measurement battery; comorbid CUD & AUD; single dose; for DTI, Bayesian parameter estimates of variance in the simple effects may be underestimated; generalizability of pioglitazone to other substances of abuse unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes